CLINICAL TRIAL: NCT04483596
Title: Efficacy of Prophylactic Melatonin to Decrease the Incidence of Postoperative Delirium in Geriatric Patients Undergoing Surgeries Under General Anesthesia. A Randomized Controlled Trial.
Brief Title: Melatonin to Decrease the Incidence of Postoperative Delirium in Geriatric Patients
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherif Abdullah Mohamed, Principal Investigator, Cairo University
Other Study IDs: MS-103-2020
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Postoperative Delirium
Keywords: melatonin; delirium; geriatrics; general anesthesia
MeSH Terms: conditions — Emergence Delirium; Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- M: will receive 5 mg melatonin orally at 9 p.m. the night before surgery and another 5 mg melatonin with 15 ml of plain water 30 min before operation and 5 mg melatonin at 9 p.m. in the day of operation and for the first three postoperative days
  Interventions: Drug: melatonin effect on the Abbreviated Mental Test
- C: received a placebo in the form of one tablet of 500 mg paracetamol that packaged the same way as melatonin at the same times
  Interventions: Drug: melatonin effect on the Abbreviated Mental Test

INTERVENTIONS:
Drug: melatonin effect on the Abbreviated Mental Test — Questionnare
  1. Age
  2. Time (to nearest hour)
  3. Address for recall at end of test (Ask patient to repeat the address to ensure it has been heard correctly)
  4. Year
  5. Name of hospital
  6. Recognition of two persons (e.g. doctor, nurse)
  7. Date of birth
  8. Year of any famous event e.g: the last Egyptian revolution
  9. Name of the present monarch
  10. Count backwards from 20 to 1

SUMMARY:
POD has been reported to be associated with a large number of risk factors: age as POD occurs in 10% to 61% of those aged 65 or older, dementia, impaired left ventricular function, electrolyte disorder, alcoholism, smoking, high perioperative transfusion requirements, intraoperative pressure fluctuation, and use of benzodiazepine POD occurs mostly in some types of surgery, such as orthopedic surgeries, major gastrointestinal surgery, and major cardiovascular surgeries, surgery under general anesthesia, prolonged surgery, emergency surgery

Previous studies done before to prove the efficacy of melatonin to decrease the incidence of postoperative delirium in patients with multiple risk factors for POD as traumatic geriatric patients were concerned only with the type of surgery as hip replacement or with spinal anesthesia but no study was done before to assess the prophylactic effect of melatonin to decrease the incidence of postoperative delirium in geriatric patients under general anesthesia ,which represents an independent risk factor for POD. So,this double blinded RCT will try to fill this gap in literature.

DETAILED DESCRIPTION:
POD has been reported to be associated with a large number of risk factors: age as POD occurs in 10% to 61% of those aged 65 or older, dementia, impaired left ventricular function, electrolyte disorder, alcoholism, smoking, high perioperative transfusion requirements, intraoperative pressure fluctuation, and use of benzodiazepine POD occurs mostly in some types of surgery, such as orthopedic surgeries, major gastrointestinal surgery, and major cardiovascular surgeries, surgery under general anesthesia, prolonged surgery, emergency surgery

Previous studies done before to prove the efficacy of melatonin to decrease the incidence of postoperative delirium in patients with multiple risk factors for POD as traumatic geriatric patients were concerned only with the type of surgery as hip replacement or with spinal anesthesia but no study was done before to assess the prophylactic effect of melatonin to decrease the incidence of postoperative delirium in geriatric patients under general anesthesia ,which represents an independent risk factor for POD. So,this double blinded RCT will try to fill this gap in literature.

Aim of the study:

To prove the efficacy of melatonin to decrease the incidence of postoperative delirium after surgeries under general anesthesia in geriatric patients.

Methodology After approval of the Research Ethics Committee and written informed consent from all patients, A randomized, prospective, controlled, double blind study of the prophylactic effect of melatonin on postoperative delirium in geriatric patients undergoing surgeries under general anesthesia will be conducted on 100 patients allocated into 2 equal groups. The study will be conducted at Cairo University Hospitals, in all surgical units.

Randomization: Patients who meet all the inclusion criteria will be randomized to either Group M (Melatonin group) or Group C (Control group) by using computer generated random numbers with closed sealed envelope.

All patients will fast according to standard rules and will be assessed by an anesthesiologist at the night before the surgery.

All patients will be screened at that time by Abbreviated Mental Test (AMT) ,where patients having scores < 6 will be considered to have postoperative delirium.This test has been recommended for routine assessment of cognitive function in the elderly by the Royal College of Physicians and the British Geriatric Society.

Questionnare (score) Each scores one point

1. Age
2. Time (to nearest hour)
3. Address for recall at end of test (Ask patient to repeat the address to ensure it has been heard correctly)
4. Year
5. Name of hospital
6. Recognition of two persons (e.g. doctor, nurse)
7. Date of birth
8. Year of any famous event e.g: the last Egyptian revolution
9. Name of the present monarch
10. Count backwards from 20 to 1

Group M (Melatonin group): will receive 5 mg melatonin orally at 9 p.m. the night before surgery and another 5 mg melatonin with 15 ml of plain water 30 min before operation and 5 mg melatonin at 9 p.m. in the day of operation and for the first three postoperative days.

Group C (Control group): received a placebo in the form of one tablet of 500 mg paracetamol that packaged the same way as melatonin at the same times.

The anesthesia residents who will administer the drug and assess Abbreviated Mental Test(AMT) score postoperatively will be blinded to the allocation regimen.

On arrival to the preparation room, wide bore IV cannula will be inserted in the nondominant hand, sedation will be assessed by Ramsay sedation scale,with grades from 1 to 6 where:1-Patient awake, anxious, agitated, or restless ,2- Patient awake, cooperative, orientated, and tranquil ,3- Patient drowsy, with response to commands ,4- Patient asleep, brisk response to glabella tap or loud auditory stimulus ,5- Patient asleep, sluggish response to stimulus ,6- Patient has no response to firm nail-bed pressure or other noxious stimuli. patients with score > 4 will be excluded from the study.

All Patients will be monitored with five lead ECG, noninvasive blood pressure, oxygen saturation, capnography and baseline HR,SBP,DBP,MAP,oxygen saturation,ETCO2 , and urine output will be recorded then every 10 minutes until 30 minutes postextubation. Induction of anesthesia will be done with fentanyl (2 mic/kg), propofol (1-2 mg/kg), atracurium (0.5 mg/kg). Intubation will be done with oral cuffed endotracheal tube size 6.5-7 mm ID for females and 7.5-8 mm ID for males and then a urinary catheter will be inserted. Anesthesia will be maintained with isoflurane (0.75- 1.15%), incremental doses of atracurium every 20 minutes and 1 mic/kg fentanyl IV if HR and/or BP increased 20% or more from baseline in response to surgical stimulation.

After surgery, patients will be transferred to PACU. Abbreviated Mental Test (AMT) scores will be reported after recovery from anesthesia (PACU AMT) and in the same day 6 hours after operation (Day-0) and in the following three postoperative days (Day-1, Day-2 and Day-3) at the same hour of assessment in day 0. Patients having scores < 6 will be considered to have postoperative delirium, and will be assessed by a psychiatrist for further management.

Postoperative pain will be managed by IV 1g paracetamol every 6 hours and 50 mg diclofenac sodium oral every 12 hours with rescue analgesia of IV nalbuphine with 0.25 mg/kg not exceeding 0.5 mg/kg every 6 hours when the numerical rating score (NRS) or advanced dementia scale (PAINAD)(if the patient developed delirium) >4.NRS or PAINAD will be evaluated according to at times 0-30 minutes 2, 4,8, 12, 18 and 24 hours. The "zero" point of time will be the moment the patient recovered from general anesthesia

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II

Exclusion Criteria:

* ASA physical status ≥ III.
* Allergy to the study drugs or one of their ingredients
* Patients with Abbreviated Mental Test (AMT) score of< 6 ,
* illiterate people,
* preoperative sedation score >4,
* History of alcohol abuse,
* Sensory impairment (blindness, deafness),
* Severe anemia (hematocrit<27%),
* Intracranial events (stroke, bleeding, infection),
* Fluid or electrolyte disturbances including dehydration, hyponatremia, hypernatremia,
* Acute cardiac events: myocardial infarction, congestive heart failure exacerbation, arrhythmia,
* Acute pulmonary events: asthma or chronic obstructive pulmonary disease exacerbation, pulmonary embolism, hypoxemia, hypercarbia -,Medications Anticonvulsants, Antidepressants, Antihistamines, Antiparkinsonian agents, Antipsychotics. And history of chronic sedative hypnotic use >3 times/week during a month prior to surgery

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: geriatric patients undergoing surgeries under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-03 (Actual)

PRIMARY OUTCOMES:
postoperative delirium | 3 postoperative days
  Detection of the difference in incidence of POD between melatonin group and control group using the Abbreviated Mental Test (AMT)

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University hospitals, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: No
not to share

REFERENCES:
- [Background] Jankowski CJ, Trenerry MR, Cook DJ, Buenvenida SL, Stevens SR, Schroeder DR, Warner DO. Cognitive and functional predictors and sequelae of postoperative delirium in elderly patients undergoing elective joint arthroplasty. Anesth Analg. 2011 May;112(5):1186-93. doi: 10.1213/ANE.0b013e318211501b. Epub 2011 Mar 17. PMID 21415433